CLINICAL TRIAL: NCT02567669
Title: Muscle Loss and Fatigue as a Consequence of Radiotherapy
Acronym: MUSFAT
Status: Active, not recruiting | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Sponsor
Other Study IDs: 008778
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Fatigue; Sarcopenia
Keywords: radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: standard postoperative radiotherapy for breast cancer — subjects will undergo ct scans to assess muscle mass and questionnaires to assess fatigue at 4 defined time points during and after radiotherapy

SUMMARY:
This study examines the extent of systemic muscle loss and the degree of fatigue experienced by breast cancer patients undergoing radiotherapy. This study seeks to identify whether muscle loss occurs outside the radiation fields and if muscle loss is correlated with the degree of fatigue.

DETAILED DESCRIPTION:
This study uses a patient reported survey to assess fatigue prior to radiotherapy for breast cancer. Fatigue is measured again at the completion of radiation treatments and at one and three months following completion of radiation.

Muscle measurements are made outside the treatment area using ct scans prior to radiation treatment, at the completion of radiation treatment and at one and three months after radiation treatment. The degree of fatigue and changes in muscle will be assessed. Changes will be correlated to determine if muscle loss contributes to fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Women Age ≥ 18 years
2. Non-metastatic breast cancer for which post-operative radiation treatment has been recommended as standard of care
3. Able to provide informed consent
4. Able to complete the Brief Fatigue Inventory questionnaire -

Exclusion Criteria:

1. Pregnant
2. Inability to meet eligibility requirements -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nonmetastatic breast cancer with indications for postoperative radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in self-reported fatigue using the validated questionnaire "Brief Fatigue Inventory" | 5 months
  Subjects will complete the Brief Fatigue Inventory questionnaire on the first day of radiation treatment, the last day of radiation treatment and one month and three months after the last radiation treatment. All dates are +/- one week. The length of radiation treatment will be determined by the treating physician as standard of care, typically four to six weeks depending on disease characteristics.
Changes in muscle area outside the radiation treatment area determined on cross sectional anatomy from CT scan images | 5 months
  Subjects will undergo ct scan imaging on the first day of radiation treatment, the last day of radiation treatment and one month and three months after the last radiation treatment. All dates are +/- one week. The length of radiation treatment will be determined by the treating physician as standard of care, typically four to six weeks depending on disease and patient characteristics. Muscle area will be determined on specified anatomic levels using automated image analysis of CT images.
Correlation between muscle area and fatigue | 5 months
  Changes in cross-sectional muscle area during and after radiotherapy will be compared with changes in self reported fatigue to determine if correlations exist between changes in fatigue and cross sectional muscle area.

SECONDARY OUTCOMES:
Changes in cross-sectional muscle area within the radiation treatment area measured on ct scans | 5 months
  cross sectional muscle area within the radiation treatment area will be measured on ct scan images at anatomic levels corresponding to irradiated tissue. changes in muscle area over the course of treatment and following treatment will be determined. muscle area will be measured on the first day of radiation treatment, the last day of radiation treatment and at one month and three months after the last radiation treatment with ct scans at all four timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Dornfeld, MD PhD, Principal Investigator — Essentia Health

IPD SHARING:
Plan to Share IPD: Yes
meeting presentation and publication